CLINICAL TRIAL: NCT04108884
Title: RedStroke - Reducing Europe's Stroke Incidence: Highly Cost-effective Population Screening Programs for Atrial Fibrillation Coupled With High Diagnostic Yield Confirmation Services
Brief Title: RedStroke - Reducing Europe's Stroke Incidence
Acronym: RedStroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: European Union (Other); Preventicus GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 2019-00908
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Smartphone App; CHA2DS2-VASc-Score; Screening; Cardiovascular risk factors; Outpatient setting; Congestive heart failure; Stroke; Diabetes; Vascular disease
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure; Stroke; Diabetes Mellitus; Vascular Diseases | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Intervention Model Description: In this study, the effect of a smartphone application in detecting AF will be assessed in a double-blind randomised controlled trial. Patients will be randomized to an intervention arm (app group) and to a standard-of-care arm (control group). Both groups will have the app installed on their private smartphones and will be asked to perform a predefined measurement protocol. The only difference between the two groups will be, that patients in the "app" group will be informed by their local PI, if the recordings of the app indicate AF, whereas the patients in the "usual care" group will obtain the read out of the app at the end of the study (6 months after inclusion).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients and study team will remain blind to the assigned groups until the end of the trial. Only in case of a positive app finding, patients and site team will be unblinded for the remaining time of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Group (Experimental): In the app group, if an episode of arrhythmia is detected with the app, the local investigator will contact the respective patient to schedule an appointment for a 14 day Holter ECG.
  Interventions: Device: App measurement; Device: 14 day Holter ECG
- Standard Care Group (Other): The control group will perform the same measurements as the intervention group, with the only difference that a cumulated Portable Document Format (PDF) report is provided after 6 months instead of the immediate feedback in the app group.
  Interventions: Device: App measurement

INTERVENTIONS:
Device: App measurement — App measurement twice a day in the first two weeks after enrollment and twice a week (on different days) from the third week onward and whenever patients feel palpitations
Device: 14 day Holter ECG — 14 day moblie patch Holter ECG for AF confirmation
  Arms: App Group

SUMMARY:
In the RedStroke study, the effect of a smartphone application in detecting Atrial Fibrillation (AF) will be assessed in a double-blind randomised controlled multicenter trial. Outpatients with an elevated risk for atrial fibrillation will be randomized to an intervention arm (app group) and to a standard-of-care arm (control group). Both groups will have the app installed on their private smartphones and will be asked to perform a predefined measurement protocol. All patients will continue their prior therapy with their general practitioner and obtain every medical treatment indicated. This study will not cause any restrictions on the usual treatment of the study patients.

The only difference between the two groups will be, that patients in the app group will be informed by their local PI, if the recordings of the app indicate AF (and obtain a 14 day Holter ECG for AF verification), whereas the patients in the "usual care" group will obtain the read out of the app at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* CHA2DS2-VASc score of 3 and above, if patients are aged under 65 years
* CHA2DS2-VASc score of 2 and above, if patients are aged 65 years or older

Exclusion Criteria:

* history of Atrial Fibrillation
* current anticoagulation treatment,
* cardiac implanted electronic device (ICD or/and PM)
* app cannot be installed due to technical problems (smartphone type, reduced smartphone storage capacity, other)
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* enrollment of the investigator, his/her family members, employees and other dependent persons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1019 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Prevalence of Atrial Fibrillation | 6 months
  Prevalence of Atrial Fibrillation confirmed by ECG in the app group compared with the standard care group

SECONDARY OUTCOMES:
Costs related to the AF screening | 6 months
  Health care resource utilization data related to AF diagnosis will be collected for all patients during the study. To evaluate the clinical consequences associated with screening, additional endpoints include the initiation of AF-related therapies including anticoagulants, antiarrhythmic agents or hospitalizations with a primary diagnosis of AF. As a general measure of health care utilization, hospitalization for any cause will also be evaluated.
Compliance of patients using the app | 6 months
  Number of patients who regularly use the app according to study instructions

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, MD, PhD, Study Director — University Hospital, Basel, Switzerland
Locations (7):
- Germany (2):
  - University Medicine Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Ambulantes Herz-Kreislauf-Zentrum, Pasewalk
- Asklepeion Hospital, Athens, Attica, Greece
- Semmelweis University - Heart and Vascular Center, Budapest, Hungary
- University Maastricht Polikliniek Hart+Vaat Centrum, Maastricht, Limburg, Netherlands
- Jagiellonian University Medical College, Krakow, Lesser Poland Voivodeship, Poland
- Universitiy Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No